CLINICAL TRIAL: NCT00798720
Title: Phase II Study of Vorinostat (SAHA, Zolinza) and Bortezomib (PS341, Velcade) as Third-Line Treatment in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Vorinostat and Bortezomib as Third-line Treatment in Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO08502; H-2008-0229 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); NCI-2011-00811 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2016-09

CONDITIONS: Carcinoma, Non Small Cell Lung
Keywords: non small cell lung cancer; HDAC; proteasome inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vorinostat + Bortezomib (Experimental): Vorinostat 400 mg + Bortezomib 1.3 mg/m2
  Interventions: Drug: vorinostat; Drug: bortezomib

INTERVENTIONS:
Drug: vorinostat — 400 mg by mouth once daily for days 1-14 of each 21 day cycle
  Other Names: SAHA; Zolinza
Drug: bortezomib — 1.3 mg/m2 IV on days 1, 4, 8, 11 of each 21 day cycle
  Other Names: PS341; Velcade

SUMMARY:
The purpose of this study is to evaluate the efficacy of vorinostat and bortezomib in the third line treatment of advanced NSCLC, as well as to assess toxicity (including neuropathy) and tolerability of this regimen.

DETAILED DESCRIPTION:
Current treatment for non-small cell lung cancer (NSCLC) remains inadequate. Vorinostat is a novel agent that inhibits the enzymatic activity of histone deacetylases (HDACs). Bortezomib is a small molecule proteasome inhibitor. Preclinical and clinical studies have shown the advantages of combining these two agents in the treatment of NSCLC

ELIGIBILITY:
Inclusion Criteria:

* Pathologically/histologically confirmed NSCLC
* Advance NSCLC (stage IIIB w/ effusion, stage IV, or recurrent disease)
* Measurable disease
* Two prior systemic anti-cancer (cytotoxic or biologic) regimens for advanced/metastatic disease, including one (1) platinum-based chemotherapy
* Prior treatment allowed if side effects have resolved and 3 weeks has passed since last dose of treatment (1 week for palliative radiation therapy)
* ECOG performance status 0, 1, or 2
* Patients with brain metastases are allowed, if clinically stable after treatment
* Normal liver, kidney, and marrow function
* 18 years of age or older
* Negative pregnancy test for women of child-bearing potential.
* Life expectancy 3 months or more
* No concurrent use of other antitumor agents

Exclusion Criteria:

* Prior therapy with vorinostat, HDAC inhibitors, or bortezomib
* Pre-existing neuropathy grade >/= 2
* Myocardial infarction within 6 months prior to enrollment or have NY Heart Association Class III or Class IV heart failure
* Have taken valproic acid </= 4 weeks prior to enrollment
* Previous or current malignancies of other histologies within the past 5 years, except cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
* Hypersensitivity to bortezomib, boron, or mannitol
* Serious medical or psychiatric illness likely to interfere with participation in the clinical study
* Pregnant women
* HIV positive patients
* Hepatitis infection (HCV or HBV) patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tien Hoang, M.D., Principal Investigator — University of Wisconsin, Madison

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred during 2/16/2008 and 03/09/2010.
Period: Overall Study
Arm/Group | Vorinostat + Bortezomib
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 57 [45 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
Histology [Number; unit: participants]
  Adenocarcinoma | 9
  Squamous Cell | 2
  NSCLC, NOS | 7
Performance Status [Number; unit: participants] — Assigned following the Eastern Cooperative Oncology Group (ECOG) scale. Scores range from 0 (fully active) to 5 (dead).
  participants
    0 | 5
    1 | 12
    2 | 1
Disease Stage [Number; unit: participants] — Disease stage per American Joint Committee on Cancer (AJCC) Lung Cancer Staging
  participants
    Metastatic | 16
    Recurrent | 2
    Brain Metastases | 6
Prior first-line systemic therapy [Number; unit: participants]
  Paclitaxel/Platinum | 10
  Paclitaxel/Platinum/Bevacizumab | 2
  Paclitaxel/Platinum/Investigational Drug | 2
  Pemetrexed/Platinum | 3
  Vinorelbine/Platinum | 1
Response to first-line therapy [Number; unit: participants]
  Partial response | 7
  Stable disease | 4
  Progressive disease | 6
  Not reported | 1
Prior second-line systemic therapy [Number; unit: participants]
  Pemetrexed | 10
  Pemetrexed/Investigational drug | 1
  Docetaxel/Investigational drug | 1
  Erlotinib | 4
  Platinum doublets | 2
Response to second-line therapy [Number; unit: participants]
  Partial response | 1
  Stable disease | 3
  Progressive disease | 13
  Not reported | 1
Prior thoracic radiation therapy [Number; unit: participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Three-month Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since the treatment started or the appearance of one or more new lesions."
Time Frame: Three-months post-treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 18
percentage of participants | 11.1 [0.8 to 25.6]

2. Secondary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) for target lesions and assessed by MRI, CT, or chest x-ray: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR+PR.
Time Frame: Until disease progression, up to 2 years
Measure: Number; unit: participants
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 18
participants
  Partial response | 0
  Stable disease | 5
  Progressive disease | 13

3. Secondary Outcome: Median Overall Survival
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 18
months | 4.7 [3.2 to 8.6]

4. Secondary Outcome: Toxicity
Description: Graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0
Time Frame: 30 days post-treatment
Measure: Number; unit: participants
Arm/Group | Vorinostat + Bortezomib
Number analyzed (Participants) | 18
participants
  Thrombocytopenia Grade 3 | 7
  Thrombocytopenia Grade 4 | 1
  Lymphopenia Grade 3 | 3
  Fatigue Grade 3 | 4
  Fatigue Grade 4 | 1
  Vomiting Grade 3 | 2
  Dizziness Grade 3 | 2
  Syncope Grade 3 | 2
  Neuropathy Grade 3 | 2
  Hyponatremia Grade 3 | 3

ADVERSE EVENTS:
Arm/Group | Vorinostat + Bortezomib
Serious Adverse Events (participants affected / at risk) | 8/18
Other Adverse Events (participants affected / at risk) | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat + Bortezomib (N=18)
Lymphopenia (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Failure to thrive (General disorders) | 1
Fatigue (General disorders) | 1
Fistula, esophagus (Gastrointestinal disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Confusion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Neuropathy, motor (Nervous system disorders) | 1
Psychosis (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes